CLINICAL TRIAL: NCT05686629
Title: A Study to Assess the Efficacy and Safety of Jaktinib Hydrochloride Tablets in the Treatment of Severe Novel Coronavirus Pneumonia
Brief Title: An Efficacy and Safety Study of Jaktinib Hydrochloride Tablets in the Treatment of Severe Novel Coronavirus Pneumonia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGJAK-IIT-004
Record Dates: First submitted 2023-01-08; First posted 2023-01-17 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Novel COVID-19-Infected Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jaktinib 100mg BID (Experimental): Jaktinib hydrochloride tablets, 2 x 50mg dosage, BID
  Interventions: Drug: Jaktinib hydrochloride tablets
- Placebo (Placebo Comparator): 2 x Placebo tablets, BID
  Interventions: Drug: Jaktinib hydrochloride tablets

INTERVENTIONS:
Drug: Jaktinib hydrochloride tablets — 2 doses per day, each containing two 50mg Jaktinib or placebo tablets

SUMMARY:
This study adopts a randomized, double-blind, placebo parallel control design, and is expected to include 120 eligible patients with severe novel coronavirus pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years old (including threshold), regardless of gender;
* There is a history of novel coronavirus antigen- or nucleic acid-positive infection within 1 week;
* HRCT is consistent with the manifestation of viral pneumonia (judged by the investigator)
* Participants who voluntarily sign informed consent.

Exclusion Criteria:

* Participants who cannot take orally, or are suspected to be allergic to Jaktinib hydrochloride, similar drugs or their excipients, or have severe gastrointestinal dysfunction that affects drug absorption;
* Critical pneumonia patients with other organ failure requiring ICU monitoring and treatment;
* Participants who have received the following treatments within the specified time window before randomization:

  1. participants have received Janus kinase (JAK) inhibitor, interleukin 6 (IL-6) inhibitor, IL-1 inhibitor, tumor necrosis factor (TNF) inhibitor, T cell or B cell depletion agent, interferon and other immunosuppressive drugs within the first two weeks of randomization, except glucocorticoid;
  2. Systematically used CYP 3A4 potent inhibitor or potent inducer in the first five drug half lives at random;
* Immune deficiency;
* Participants who have received novel coronavirus vaccine within 1 week before randomization;
* Prior to randomization, there were the following active and uncontrolled infections: tuberculosis, HIV, syphilis, mycoplasma, chlamydia, parasites, and viral infections other than SARS CoV-2 that required systemic anti-infection treatment;
* Renal diseases requiring dialysis treatment;
* Pregnant and lactating women;
* Any other participants that were considered unsuitable by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Jaktinib | 14 days after randomization
  The proportion of subjects with disease progression or all-cause mortality;
Efficacy of Jaktinib | 28 days after randomization
  The proportion of subjects with disease progression or all-cause mortality;
Efficacy of Jaktinib | 28 days after randomization
  The proportion of subjects whose (National Institute of Allergy and Infectious Disease Ordinal Scale (NIAID-OS) score improved by ≥ 2 points from the baseline
Efficacy of Jaktinib | 28 days after randomization
  The change value of NIAID-OS score compared with the baseline
Efficacy of Jaktinib | up to 28 days after randomization
  Time interval from randomization to clinical improvement (defined as NIAID-OS 1-3 points)
Time interval from randomization to discharge | up to 28 days after randomization
Efficacy of Jaktinib | 28 days after randomization
  The proportion of subjects receiving mechanical ventilation due to disease progression at 3, 7, 14 days after randomization until end of treatment (EOT)
Efficacy of Jaktinib | 28 days after randomization
  the proportion of subjects whose chest High-Resolution CT (HRCT) showed significant absorption of pulmonary inflammation (definition of significant absorption: the lung inflammatory lesions were reduced by more than 50%) at 7, 14 days after treatment until EOT

SECONDARY OUTCOMES:
Safety of Jaktinib | up to 2 months after randomization
  Incidence rate of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Li, Prof., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No